CLINICAL TRIAL: NCT07318779
Title: Effect of Cardamom and Peppermint Oils on Chemotherapy-Related Nausea-Vomiting and Food Intake: Randomized Controlled Study
Brief Title: Effect of Cardamom and Peppermint Oils on Chemotherapy-Related Nausea-Vomiting and Food Intake
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semanur Bilgiç (Other)
Responsible Party: Sponsor-Investigator, Semanur Bilgiç, Research Assistant, Bilecik Seyh Edebali Universitesi
Organization: Bilecik Seyh Edebali Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Chemotherapy
Record Dates: First submitted 2025-11-19; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Aromatherapy; Chemotherapy; Nausea; Vomiting; Food Intake
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting | interventions — peppermint oil; almond oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- peppermint oil (Experimental): Thirty minutes before the chemotherapy session begins, one drop of essential oil will be applied to a piece of gauze. The gauze will then be attached to the patient's collar with a safety pin, positioned 20 cm away from the patient's nose. This procedure will be performed three times a day for five consecutive days.
  Interventions: Other: Peppermint Oil
- cardamom oil (Active Comparator): Thirty minutes before the chemotherapy session begins, one drop of essential oil will be applied to a piece of gauze. The gauze will then be attached to the patient's collar with a safety pin, positioned 20 cm away from the patient's nose. This procedure will be performed three times a day for five consecutive days.
  Interventions: Other: cardomom oil
- sweet almond oil (Sham Comparator): Thirty minutes before the chemotherapy session begins, one drop of essential oil will be applied to a piece of gauze. The gauze will then be attached to the patient's collar with a safety pin, positioned 20 cm away from the patient's nose. This procedure will be performed three times a day for five consecutive days.
  Interventions: Other: sweet almond oil

INTERVENTIONS:
Other: Peppermint Oil — Thirty minutes before the chemotherapy session begins, one drop of essential oil will be applied to a piece of gauze. The gauze will then be attached to the patient's collar with a safety pin, positioned 20 cm away from the patient's nose. This procedure will be performed three times a day for five consecutive days.
  Arms: peppermint oil
Other: cardomom oil — Thirty minutes before the chemotherapy session begins, one drop of essential oil will be applied to a piece of gauze. The gauze will then be attached to the patient's collar with a safety pin, positioned 20 cm away from the patient's nose. This procedure will be performed three times a day for five consecutive days.
  Arms: cardamom oil
Other: sweet almond oil — Thirty minutes before the chemotherapy session begins, one drop of essential oil will be applied to a piece of gauze. The gauze will then be attached to the patient's collar with a safety pin, positioned 20 cm away from the patient's nose. This procedure will be performed three times a day for five consecutive days.
  Arms: sweet almond oil

SUMMARY:
The aim of this study is to evaluate the effect of inhaled cardamom oil on chemotherapy-related nausea, vomiting, and food intake and to compare these effects with those of inhaled peppermint oil.

DETAILED DESCRIPTION:
Chemotherapy is an effective treatment method used to control cancer systemically by destroying cancer cells or controlling their growth. This treatment inhibits nucleic acid synthesis, thereby preventing DNA and RNA synthesis, and has both cytotoxic and anticancer properties. However, chemotherapy also affects rapidly dividing cells, leading to undesirable side effects. Among these, nausea and vomiting are common and quality-of-life-reducing side effects that affect approximately 80% of patients undergoing chemotherapy.

The pathophysiology of nausea and vomiting is based on mechanisms such as the stimulation of the vomiting center and the chemoreceptor trigger zone, as well as the stimulation of enterochromaffin cells and vagal afferent neurons. Failure to manage these symptoms can lead to serious problems such as malnutrition, dehydration, anorexia, and fluid-electrolyte imbalance. Therefore, antiemetic drugs and various integrative methods (acupuncture, acupressure, behavioral interventions, music therapy, relaxation exercises, hypnotherapy, and aromatherapy) are used to manage nausea and vomiting.

Aromatherapy with various essential oils such as peppermint, ginger, rose, cardamom, lavender, and chamomile has been found to be effective in preventing nausea and vomiting. The effect of peppermint oil on chemotherapy-related nausea and vomiting is well-documented; however, research on cardamom oil is limited. There are few studies in the literature evaluating the effect of cardamom oil on these symptoms. The aim of this study is to evaluate the effect of inhaled cardamom oil on chemotherapy-related nausea, vomiting, and food intake and to compare these effects with those of inhaled peppermint oil.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study,
* Received at least one cycle and are continuing to receive either Adriamycin-cyclophosphamide or Adriamycin-cyclophosphamide-fluorouracil chemotherapy protocols,
* Have an intact sense of smell.

Exclusion Criteria:

* Under 18 years of age,
* Have neurocognitive impairment and are unable to answer the questionnaire,
* Have a condition that may trigger nausea and vomiting, such as vertigo or motion sickness,
* Have a chronic respiratory disease (with a history of asthma or other reactive airway diseases),
* Have a known history of allergies,
* Have a history of prolonged or excessive alcohol use,
* Use any scented products during the intervention period,
* Receive other complementary therapies for nausea and vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-Related Nausea-Vomiting and Retching | five consecutive days.
  The Rhodes Index of Nausea, Vomiting and Retching (INVR) was developed by Rhodes and McDaniel in 1999 to assess nausea, vomiting, retching, and related distress experienced within the last 12 hours, particularly after chemotherapy. The scale consists of 8 items rated on a Likert-type scale, where 0 indicates minimal distress and 4 indicates severe distress. Items 1, 3, 6, and 7 are reverse-scored. The INVR includes three subdimensions: symptom experience, symptom occurrence, and symptom distress. The original scale demonstrated high internal consistency (Cronbach's alpha = 0.98; subscales = 0.83-0.99).
Food Intake | five consecutive days.
  Food Consumption Form:
  The 24-hour dietary recall method is used to record food intake. In this study, patients record all foods and beverages consumed over five consecutive days. Portions are documented using household measures such as cups, glasses, mugs, and spoons.
Chemotherapy-Related Nausea | five consecutive days.
  Visual Analog Scale (VAS):
  The severity of nausea will be assessed using a 100-mm Visual Analog Scale (VAS), where the left end represents "no nausea" and the right end represents "severe nausea." A score <5 mm is defined as no nausea, and a 10-mm difference is typically considered clinically significant.
Food Frequency Form | five consecutive days.
  This form identifies the food groups consumed by the patient over the five-day period. It verifies the information recorded in the food consumption form and provides insight into the patient's dietary patterns. The food frequency method is commonly used to assess relationships between diet and disease risk.
Anthropometric Measurements1 | Measurements will be taken twice, on the first and fifth days.
  Body mass index (BMI) is calculated by dividing weight in kilograms by height in meters squared (kg/height²).
Anthropometric Measurements2 | Measurements will be taken twice, on the first and fifth days.
  Skinfold thickness measurements are taken using calipers and are used to rank individuals in terms of relative total "fatness" or to assess subcutaneous fat in various areas of the body.
Anthropometric Measurements3 | Measurements will be taken twice, on the first and fifth days.
  waist and hip circumference: Using a tape measure, measure around the narrowest part of the waist, just above the belly button. This is the waist circumference. Measure around the widest part of the hips. This is the hip circumference.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir City Hospital, Eskişehir, Turkey (Türkiye)